CLINICAL TRIAL: NCT00807027
Title: Multi-center, Randomized, Open-label Phase 3 Clinical Trial to Assess the Efficacy and Safety of 'INNOCELL Immuncell-LC' With Temozolomide in Newly Diagnosed Glioblastoma of Korea
Brief Title: Clinical Trial to Assess the Efficacy and Safety of 'Immuncell-LC' With Temozolomide in Newly Diagnosed Glioblastoma of Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IcmLCBT_301
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Newly diagnosed Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): The study subjects randomly assigned to the control group is given Temozolomide chemotherapy and radiation therapy for 6 weeks according to the clinical test plans, and then administers Temozolomide only for 6 weeks.
- Test Group (Experimental): The study subjects assigned to the test group blood is drawn before minimum 2 weeks in order to manufacture the test drug. Test group is compared its progression free survival rate after surgery by administering Temozolomide chemotherapy and radiation therapy same as control group with Immuncell-LC (14 times).
  Interventions: Drug: Activated T lymphocyte(Immuncell-LC)

INTERVENTIONS:
Drug: Activated T lymphocyte(Immuncell-LC) — Efficacy/Effects: Removal of minimal residual cancer after removal of brain tumors and relapse prevention
  Method of administration and quantity: Test Drug: Per 60kg of average adult body weight, administer 100mg that contains 109~2x1010 lymphocytes for one hour intravenously. (Duration of administration can be controlled based on patient conditions)
  Arms: Test Group

SUMMARY:
This clinical study was planned in order to assess the superiority of INNOCELL Corp. "Immuncell-LC" in aspects of therapeutic efficacy and safety when administered with Temozolomide to glioblastoma patients when compared with the control group who did not receive administration of the drug.

DETAILED DESCRIPTION:
<Primary Purpose> Compare clinical efficacy of group treated with cell theraputic INNOCELL Immuncell-LC evaluated by progression free survival with that of untreated group.

<Secondary Purpose> Compare clinical efficacy of group treated with INNOCELL Immuncell-LC, a drug for treating glioblastoma evaluated by overall survival, therapy reaction, EORTC QLQ-C30, and Karnofsky Performance Status (KPS) and that of untreated group, and evaluate adverse reactions, clinical pathological tests, and its safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who, prior to the study, received explanation of the purpose and content of study and of characteristics of the test drug from the test administrator and have consented to the study by providing signature of self, guardian, or legal representative.
2. Patients who are between 18 and 70 years of age
3. Patients whose cause of cancer has been found to be glioblastoma via pathological testing
4. patients who have received surgery for glioblastoma (Complete or partial extirpation or biopsy) 2 weeks prior to the study
5. Patients whose survival is expected to be longer than 3 months
6. Patients whose KPS is greater than 60
7. Patients who satisfy the following conditions of the blood test, kidney function test, and liver function test

   * Hemoglobin is bigger than 10 gm%
   * Platelet Count is bigger than 100,000/µL
   * Absolute granulocyte count is bigger than 1,500/µL
   * BUN or Creatinine 1.5 x upper normal limit
   * Bilirubin level is smaller than 2.0 mg/dL
   * SGOT, SGPT, alkaline phosphatase is smaller than 1.5 x upper normal limit

Exclusion Criteria:

1. Patients who have been determined to have serious Cardio - Pulmonary function disability by the clinical study staff
2. Patients who are immune deficient or have a history of auto immune diseases (Ex. Rheumatoid Arthritis, Systemic Lupus Erythematosus, Vasculitis, Multiple sclerosis, Adolescent Insulin-Dependent Diabetes Mellitus, etc.)
3. Patients who have a history of malignant tumors in the recent 5 years prior to the study with the exception of skin cancer, local prostate cancer, and cervical cancer.
4. Patients with history of severe allergies
5. Patients with serious mental illness
6. Patients who are pregnant or nursing
7. Patients who have participated in other clinical tests in the recent 4 weeks prior to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-12-05 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chunghyun Kim, MD, Principal Investigator — Hanyang University
Locations (7):
- South Korea (7):
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Gyunghee University Medical Center, Seoul
  - Konkuk University, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Seoul Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul
  - Yeonsei University Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- CIK Immunotherapy Group: The study subjects assigned to the test group blood is drawn before minimum 2 weeks in order to manufacture the test drug. Test group is compared its progression free survival rate after surgery by administering Temozolomide chemotherapy and radiation therapy same as control group with Immuncell-LC (14 times).
  Activated T lymphocyte(Immuncell-LC): Efficacy/Effects: Removal of minimal residual cancer after removal of brain tumors and relapse prevention
  Method of administration and quantity: Test Drug: Per 60kg of average adult body weight, administer 100mg that contains 109~2x1010 lymphocytes for one hour intravenously. (Duration of administration can be controlled based on patient conditions)
Period: Overall Study
Arm/Group | Control Group | CIK Immunotherapy Group
Started | 89 | 91
Completed | 73 | 74
Not Completed | 16 | 17
Not completed — Withdrawal by Subject | 13 | 14
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: From December 2008 to October 2012, a total of 188 patients were screened from 7 institutes in Korea, 8 patients failed in the screening process, and 180 patients were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | CIK Immunotherapy Group | Total
Number analyzed (Participants) | 89 | 91 | 180
Age, Continuous [Median (Full Range); unit: years] | 54.0 [23.0 to 68.0] | 55.0 [19.0 to 69.0] | 54.5 [19.0 to 69.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 51 | 51 | 102
Region of Enrollment [Number; unit: participants]
  South Korea | 89 | 91 | 180
Karnofsky performance scale [Median (Full Range); unit: units on a scale] — The Karnofsky Performance Scale (KPS) measures a patient's functional status and ability to carry out daily activities. Scores range from 0 to 100, where:
  * 100 = Normal, no complaints, no evidence of disease (best outcome)
  * 70 = Cares for self, unable to carry on normal activity or active work
  * 40 = Disabled, requires special care and assistance
  * 0 = Dead (worst outcome) Higher scores represent better functional status. Scores are reported as units on a scale.
  units on a scale | 90 [60.0 to 100.0] | 90.0 [60.0 to 100.0] | 90.0 [60.0 to 100.0]
Global health status/Quality of life [Median (Full Range); unit: units on a scale] — European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) - a validated, cancer-specific instrument designed to assess the quality of life of cancer patients. The Global Health Status/Quality of Life (QoL) scale is one of the multi-item scales included in the instrument.
  The Global Health Status/QoL scale is scored from 0 to 100. Scores are transformed linearly following the EORTC scoring manual. Higher scores represent better health status and quality of life. Lower scores indicate poorer poorer perceived health and quality of life.
  units on a scale | 50 [0.0 to 100] | 58 [8.0 to 100] | 54 [0.0 to 100]
Tumor size [Median (Full Range); unit: centimeter] | 1.4 [0.0 to 67.1] | 4.2 [0.0 to 28.2] | 2.8 [0.0 to 67.1]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival(PFS)
Description: Progression-free survival was assessed locally by investigators on the basis of enhanced MRI was performed approximately 4 weeks after chemoradiotherapy, then at 10, 22, 34 and 46 weeks after randomization, and every 3~12 months thereafter during the follow-up phase.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 46 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Control Group | CIK Immunotherapy Group
Number analyzed (Participants) | 89 | 91
months | 5.4 [3.3 to 7.9] | 8.1 [5.8 to 8.5]

2. Secondary Outcome: Overall Survival(OS)
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CIK Immunotherapy Group: The study subjects assigned to the test group blood is drawn before minimum 2 weeks in order to manufacture the test drug. Test group is compared its progression free survival rate after surgery by administering Temozolomide chemotherapy and radiation therapy same as control group with Immuncell-LC (14 times).
  Activated T lymphocyte(Immuncell-LC): Efficacy/Effects: Removal of minimal residual cancer after removal of brain tumors and relapse prevention
  Method of administration and quantity: Test Drug: Per 60kg of average adult body weight, administer 100mg that contains 10^9~2x10^10 lymphocytes for one hour intravenously. (Duration of administration can be controlled based on patient conditions)
Arm/Group | Control Group | CIK Immunotherapy Group
Number analyzed (Participants) | 89 | 91
months | 16.88 [13.91 to 21.94] | 22.47 [17.20 to 23.85]

ADVERSE EVENTS:
Groups:
- Test Group: The study subjects assigned to the test group blood is drawn before minimum 2 weeks in order to manufacture the test drug. Test group is compared its progression free survival rate after surgery by administering Temozolomide chemotherapy and radiation therapy same as control group with Immuncell-LC (14 times).
  Activated T lymphocyte(Immuncell-LC): Efficacy/Effects: Removal of minimal residual cancer after removal of brain tumors and relapse prevention
  Method of administration and quantity: Test Drug: Per 60kg of average adult body weight, administer 100mg that contains 109~2x1010 lymphocytes for one hour intravenously. (Duration of administration can be controlled based on patient conditions)
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 52/89 | 51/91
Serious Adverse Events (participants affected / at risk) | 31/89 | 35/91
Other Adverse Events (participants affected / at risk) | 83/89 | 84/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=89) | Test Group (N=91)
Convulsion (Nervous system disorders) | 3 (3) | 6 (9)
Headache (Nervous system disorders) | 5 (5) | 4 (5)
Brain edema (Nervous system disorders) | 2 (2) | 4 (4)
Hemiparesis (Nervous system disorders) | 4 (4) | 2 (2)
Hydrocephalus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Mental impairment (Nervous system disorders) | 3 (3) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
paraparesis (Nervous system disorders) | 0 (0) | 2 (2)
Partial seizure (Nervous system disorders) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
cerebral cyst (Nervous system disorders) | 0 (0) | 1 (1)
cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
somnolence (Nervous system disorders) | 1 (1) | 0 (0)
speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 4 (4) | 3 (3)
sepsis (Infections and infestations) | 0 (0) | 2 (2)
septic shock (Infections and infestations) | 1 (1) | 1 (1)
appendicitis (Infections and infestations) | 1 (1) | 0 (0)
bacteriaemia (Infections and infestations) | 1 (1) | 0 (0)
enterits infectious (Infections and infestations) | 1 (1) | 0 (0)
lung abscess (Infections and infestations) | 1 (1) | 0 (0)
meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
pyrexia (General disorders) | 2 (2) | 2 (2)
asthenia (General disorders) | 1 (1) | 2 (2)
chills (General disorders) | 1 (1) | 0 (0)
general physical health deterioration (General disorders) | 1 (1) | 0 (0)
multi-organ failure (General disorders) | 1 (1) | 0 (0)
concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
rib fracure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
subdural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pneumothroax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
platelet count decreased (Investigations) | 0 (0) | 1 (1)
white blood cell count decreased (Investigations) | 0 (0) | 1 (1)
hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=89) | Test Group (N=91)
Nausea (Gastrointestinal disorders) | 52 (90) | 46 (92)
Constipation (Gastrointestinal disorders) | 31 (40) | 32 (40)
Vomiting (Gastrointestinal disorders) | 28 (46) | 34 (65)
Dyspepsia (Gastrointestinal disorders) | 20 (28) | 16 (24)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 17 (18)
Abdominal Discomfort (Gastrointestinal disorders) | 3 (5) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 4 (8)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecal Incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum itestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 51 (51) | 51 (51)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (20) | 13 (20)
Rash (Skin and subcutaneous tissue disorders) | 8 (10) | 9 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (10)
Swelling Face (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3)
Skin Disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 29 (38) | 28 (47)
Tremor (Nervous system disorders) | 13 (15) | 15 (18)
Convulsion (Nervous system disorders) | 12 (16) | 15 (21)
Hemiparesis (Nervous system disorders) | 12 (15) | 11 (14)
Dizziness (Nervous system disorders) | 13 (17) | 7 (8)
Brain oedema (Nervous system disorders) | 6 (6) | 11 (11)
Mental impairment (Nervous system disorders) | 8 (11) | 9 (11)
Neuropathy peripheral (Nervous system disorders) | 6 (7) | 6 (7)
Memory impairment (Nervous system disorders) | 3 (3) | 7 (7)
Paresthesia (Nervous system disorders) | 6 (6) | 4 (4)
dysarthria (Nervous system disorders) | 3 (3) | 6 (6)
Hydrocephalus (Nervous system disorders) | 4 (4) | 4 (4)
Lethargy (Nervous system disorders) | 1 (1) | 7 (8)
Monoparesis (Nervous system disorders) | 2 (2) | 5 (5)
Somnolence (Nervous system disorders) | 4 (4) | 3 (3)
Speech disorder (Nervous system disorders) | 4 (4) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 4 (6)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 2 (2)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 4 (4)
Cognitive disorder (Nervous system disorders) | 3 (3) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 4 (4)
Partial Seizures (Nervous system disorders) | 1 (2) | 3 (3)
Aphasia (Nervous system disorders) | 0 (0) | 3 (3)
Facial paresis (Nervous system disorders) | 2 (2) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Cereral cyst (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Facial spasm (Nervous system disorders) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Head titubation (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Neurologic neglect syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 50 (74) | 54 (71)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Deydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes melitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 23 (28) | 25 (36)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 7 (7)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5)
Herpes zoster (Infections and infestations) | 2 (2) | 6 (6)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Oral candidasis (Infections and infestations) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 2 (2)
sepsis (Infections and infestations) | 0 (0) | 3 (3)
Bacteriuria (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bateraemia (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter Gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis asceptic (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
PEritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinsitis (Infections and infestations) | 0 (0) | 1 (1)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tonsllitis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 14 (20) | 27 (47)
Asthenia (General disorders) | 16 (16) | 14 (17)
Fatigue (General disorders) | 12 (13) | 15 (17)
Face oedema (General disorders) | 8 (8) | 7 (8)
Pain (General disorders) | 7 (7) | 8 (9)
Oedema peripheral (General disorders) | 2 (3) | 10 (10)
Chills (General disorders) | 3 (3) | 8 (11)
oedema (General disorders) | 4 (4) | 7 (7)
Chest discomfort (General disorders) | 4 (4) | 6 (7)
Gait disturbance (General disorders) | 2 (2) | 3 (3)
Generalised oedema (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Gait deviation (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 19 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (11) | 18 (23)
Neutrophil count decreased (Investigations) | 7 (8) | 15 (19)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 9 (10)
Platelet count decreased (Investigations) | 3 (3) | 9 (12)
White blood cell count decreased (Investigations) | 2 (3) | 8 (18)
Haemoglobin decreased (Investigations) | 2 (2) | 5 (6)
Hepatic enzyme increased (Investigations) | 4 (4) | 2 (2)
Blood sodium decreased (Investigations) | 2 (2) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Ammonia increased (Investigations) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2)
Skin test positive (Investigations) | 0 (0) | 2 (15)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Clostridium test positive (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Electocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (11)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 10 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Slep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 3 (3) | 6 (6)
Eye pain (Eye disorders) | 6 (6) | 1 (1)
Visual impairment (Eye disorders) | 3 (3) | 2 (2)
Diplopia (Eye disorders) | 3 (3) | 1 (1)
Eyelid oedema (Eye disorders) | 4 (4) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Glare (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1)
Visual activity reduced (Eye disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (13) | 13 (16)
Leukopenia (Blood and lymphatic system disorders) | 7 (8) | 16 (26)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 4 (8)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 4 (6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (9) | 8 (10)
Depression (Psychiatric disorders) | 6 (7) | 5 (5)
Mood altered (Psychiatric disorders) | 2 (2) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 5 (5) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 6 (6)
Haematuria (Renal and urinary disorders) | 1 (1) | 5 (5)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 2 (2)
Nurogenic bladder (Renal and urinary disorders) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Enurresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Rnal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 4 (5)
Ear abrasion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (3)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint disclocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 5 (6)
Flushing (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
shock (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (3) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2)
otorrhoea (Ear and labyrinth disorders) | 1 (1) | 2 (4)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Auricular swelling (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Calculus prostatic (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Galactorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 4 (4) | 1 (4)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No